CLINICAL TRIAL: NCT04701411
Title: A Phase 3, Open-Label, Multicenter Study to Evaluate the Efficacy and Safety of Darvadstrocel in the Treatment of Complex Perianal Fistula in Pediatric Subjects With Crohn's Disease Over a Period of 24 Weeks and an Extended Follow-up Period for a Total of up to 52 Weeks
Brief Title: A Study of Darvadstrocel for Treating Complex Perianal Fistulas in Children and Teenagers With Crohn's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Darvadstrocel-3004; 2020-003193-48 (EudraCT Number); EMEA-001561-PIP01-13-M02 (Other: EU PIP number); 2023-503973-39-00 (EU CTIS Number: EU CTIS Number); jRCT2033200314 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Crohn's Disease; Complex Perianal Fistula
Keywords: Drug therapy.
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Darvadstrocel (Experimental): Participants were administered darvadstrocel (Cx601), 24 milliliters (mL) suspension of 120 million cells as a perilesional injection, once on Day 0.
  Interventions: Biological: Darvadstrocel

INTERVENTIONS:
Biological: Darvadstrocel — Darvadstrocel perilesional injection.
  Other Names: Cx601

SUMMARY:
A perianal fistula is an abnormal passageway that develops between the rectum and the skin near the anus. The fistula is considered complex if it branches into several openings or an abscess is also present.

The main aim of this study is to learn if complex perianal fistulas in children and teenagers close after treatment with darvadstrocel.

2 to 3 weeks before treatment with darvadstrocel, each participant will have surgery to clean the fistula and to drain any abscesses. On the day of treatment, each participant will have the fistula cleaned and will receive an injection of darvadstrocel near the fistula, under anesthetic.

For up to 1 year after treatment, participants will regularly visit the clinic for follow-up. The fistula will be examined and any side effects from the treatment will be recorded. Participants will have an MRI at one clinic visit (about 24 weeks after treatment).

DETAILED DESCRIPTION:
The drug being tested in this study is called darvadstrocel (Cx601, cell suspension containing 120 million cells of allogeneic expanded adipose-derived mesenchymal stem cells [eASCs]). Darvadstrocel is being tested to treat complex perianal fistula in pediatric participants who have Crohn's disease (CD). This study will look at the safety and efficacy of darvadstrocel in the treatment of complex perianal fistula in CD.

The study will enroll at least 20 patients who will receive a single dose of darvadstrocel.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is 52 weeks.

Participants will make multiple visits to the clinic. In unavoidable circumstances, such as the coronavirus disease 2019 pandemic, exceptions may be granted for alternative methods for conducting participant visits with approval by the medical monitor and/or sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Has a CD diagnosis based on accepted clinical, endoscopic, histological and/or radiologic criteria at least 6 months before the screening visit.
2. Has complex perianal fistula refractory to at least one of the following treatments: immunosuppressants or biologics (anti-TNFs, anti-integrin, anti-interleukin [IL] 12/23). Fistula(s) refractory to therapy is defined in this study as follows: Immunosuppressants: Inadequate response after 3 months, based on clinical assessment, or more treatment with azathioprine, 6-mercaptopurine or methotrexate. Biologics: Inadequate response after 14 weeks (16 weeks for anti-IL 12/23), based on clinical assessment, or more standard treatment for induction and maintenance.
3. A complex perianal fistula(s) that meets one or more of the following criteria, modified from the American Gastroenterological Association (AGA) technical review: High intersphincteric, transsphincteric, extrasphincteric, or suprasphincteric as assessed by MRI. Presence of 2 or 3 external openings (tracts) as assessed by clinical examination. Associated fluid (abscess) collections as determined by MRI.

   This study requires that the participant has complex perianal fistulas with a maximum of 2 internal openings and a maximum of 3 external openings, based on clinical assessment. Darvadstrocel treatment is targeted for fistulas that connect between internal and external openings. A central reading of a locally performed pelvic MRI will be performed to confirm the location of the fistula and potential associated perianal abscess(es). Fistulas must have been draining for at least 6 weeks before the screening visit. Participants with actively draining simple subcutaneous fistulas, at the time of the screening visit, are not allowed in this study.
4. Has inactive or mildly active luminal CD defined by meeting all of the following criteria:

   1. Colonoscopy, flexible sigmoidoscopy or rectoscopy performed either at screening or within the 6 months before screening, demonstrating no rectal ulcers larger than 0.5 cm. A participant who has documented rectal ulcers larger than 0.5 cm within the 6 months before screening but has undergone subsequent treatment may be eligible if there are no rectal ulcers larger than 0.5 cm on a sigmoidoscopy or rectoscopy performed after treatment or at the time of screening.
   2. The improvement of, or no worsening in stool frequency, sustained for 1 week or more, in the interval between the colonoscopy, flexible sigmoidoscopy or rectoscopy in inclusion criteria 4(a) and the screening visit.
   3. No initiation or intensification of treatment with corticosteroids, immunosuppressants, or monoclonal antibody dose regimen between the colonoscopy, flexible sigmoidoscopy or rectoscopy in inclusion criteria 4(a) and the screening visit.

Exclusion Criteria:

1. Has received any investigational compound within 12 weeks/84 days before screening.
2. Has received darvadstrocel/eASC in a previous clinical study or as a therapeutic agent.
3. The participant weighs <10 kg at screening.
4. Has concomitant perianal fistula(s) with only internal or external opening(s).
5. Has concomitant internal fistula(s) such as ileo-vesical, rectovaginal or ileo-colonic fistula(s).
6. Has an abscess >2 cm, unless resolved in the preparation procedure.
7. Has rectal and/or anal stenosis, and/or active proctitis, which would restrict the surgical procedure.
8. The participant underwent surgery for the fistula other than drainage or seton placement.
9. Has diverting stomas.
10. Has ongoing systemic corticosteroid treatment or has been treated with systemic corticosteroids within 4 weeks before screening.
11. The participant requires new treatment with immunosuppressants/anti-TNF agents during the screening period.
12. The participant has known or suspected COVID-19 by the investigator within the past 2 months (additional testing may be performed at the discretion of the investigator). Positive antibody testing for COVID without other evidence of current or recent active infection does not exclude participation. Participants who were in screening at the time that COVID-19-related factors resulted in discontinuation may also be rescreened with approval of the sponsor or designee.
13. The participant requires surgery in the perianal region for reasons other than fistulas at the time of screening or foreseen either during the study and/or during the 24 weeks after treatment administration.
14. Has malignant tumor or a prior history of any malignant tumor, including any type of fistula carcinoma.
15. Has current or recent (within 3 months before the screening) history of abnormal, severe, progressive, uncontrolled hepatic, hematologic, gastrointestinal (except CD), endocrine, pulmonary, cardiac, neurological, psychiatric, or cerebral disease.
16. Has either congenital or acquired immunodeficiencies, including participants known to be HIV carriers or participants with, in the judgment of the investigator, are suspected to have monogenic inflammatory bowel disease.
17. Has previously received a bone marrow transplant.
18. Has a contraindication to MRI scan or other planned study procedures.
19. Has a contraindication to the anesthetic procedure.
20. Had major surgery or severe trauma within 6 months before the screening visit.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (22):
- Israel (5):
  - Shamir Medical Center (Assaf Harofeh), Be’er Ya‘aqov
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital-Mt. Scopus, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
- Japan (5):
  - Juntendo University Hospital, Bunkyō City
  - Medical Hospital, Tokyo Medical and Dental University, Bunkyō City
  - Miyagi Children's Hospital, Sendai
  - Jichi Medical University Hospital, Shimotsuke-shi
  - Mie University Hospital, Tsu
- Netherlands (3):
  - Amsterdam UMC, Locatie AMC, Amsterdam
  - Universitair Medisch Centrum Groningen (UMCG), Groningen
  - Erasmus Medisch Centrum, Rotterdam
- Poland (3):
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów
  - Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw
- Spain (6):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Materno-Infantil de Malaga, Málaga

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be reidentified (due to the limited number of study participants/study sites.

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60096520565ce300294c6adf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites globally from 30 June 2021 to 07 May 2025.
Pre-assignment Details: Participants with complex perianal fistula due to Crohn's Disease (CD) participated in this study to receive darvadstrocel (Cx601). The study was terminated early based on the sponsor's decision and did not meet the planned enrollment number. All enrolled participants completed all the study assessments.
Period: Overall Study
Arm/Group | Darvadstrocel
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received the study treatment.
Groups:
- Darvadstrocel: Participants were administered darvadstrocel (Cx601), 24 mL suspension of 120 million cells as a perilesional injection, once on Day 0.
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.7 (1.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Combined Remission
Description: Combined remission was defined as the closure of all treated external openings that were draining at baseline despite gentle finger compression, and absence of abscess(es) >2 centimeters (cm) (in at least 2 dimensions) of the treated perianal fistula(s) confirmed by central magnetic resonance imaging (MRI) assessment.
Time Frame: Week 24
Population: Intent-to-treat (ITT) analysis set included all participants who underwent the fistula preparation procedure regardless of being treated or not.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 7
percentage of participants | 42.9 [9.9 to 81.6]

2. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission
Description: Clinical remission was defined as the closure of all treated external openings that were draining at baseline despite gentle finger compression.
Time Frame: Weeks 24 and 52
Population: ITT analysis set included all participants who underwent the fistula preparation procedure regardless of being treated or not.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 7
percentage of participants
  Week 24 | 42.9 [9.9 to 81.6]
  Week 52 | 28.6 [3.7 to 71.0]

3. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response
Description: Clinical response was defined as closure of at least 50% of all treated external openings that were draining at baseline despite gentle finger compression.
Time Frame: Weeks 24 and 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 7
percentage of participants
  Week 24 | 71.4 [29.0 to 96.3]
  Week 52 | 28.6 [3.7 to 71.0]

4. Secondary Outcome: Time to Clinical Remission
Description: Time to Clinical Remission was defined as the time in weeks from treatment start to first visit at which clinical remission was observed before Week 52; where clinical remission is said to have occurred if a clinical assessment showed closure of all treated external openings that were draining at baseline despite gentle finger compression. Participants without documented time to clinical remission by the end of study (Week 52), were censored at the date of last assessment along with the participants who discontinued without clinical remission before Week 52 at the date of last visit.
Time Frame: Up to Week 52
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 7
weeks | NA [6.1 to NA] — Median and upper limit of 95% confidence interval (CI) were not estimable due to insufficient number of participants with events.

5. Secondary Outcome: Time to Clinical Response
Description: Time to clinical response defined as the time in weeks from treatment start to first visit at which clinical response was observed before Week 52; where clinical response is said to have occurred if a clinical assessment showed closure of at least 50% of all treated external openings that were draining at baseline despite gentle finger compression. Participants without documented time to clinical response by the end of study (Week 52), were censored at the date of last assessment along with the participants who discontinued without clinical response before Week 52 at the date of last visit.
Time Frame: Up to Week 52
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 7
weeks | 6.6 [6.1 to NA] — The upper limit of 95% CI was not estimable due to censoring.

6. Secondary Outcome: Percentage of Participants With Relapse in Participants With Combined Remission at Week 24
Description: Relapse was defined as reopening of any of the treated fistula(s) external openings with active drainage as clinically assessed in participants who were in combined remission at Week 24.
Time Frame: From Week 24 to Week 52
Population: ITT analysis set included all participants who underwent the fistula preparation procedure regardless of being treated or not. Overall number analyzed is the number of participants with combined remission at Week 24.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 3
percentage of participants | 0.0 [0.0 to 70.8]

7. Secondary Outcome: Percentage of Participants With At Least One Treatment-Emergent Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent AE is an AE which occurs after exposure to study treatment.
Time Frame: Up to Week 52
Population: Safety analysis set included all participants who received the study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 7
percentage of participants | 85.7

8. Secondary Outcome: Percentage of Participants With At Least One Treatment-Emergent Serious Adverse Event (SAE)
Description: An SAE is defined as an untoward medical occurrence, significant hazard, contraindication, side effect or precaution that at any dose: results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant. A treatment-emergent SAE is an SAE which occurs after exposure to study treatment.
Time Frame: Up to Week 52
Population: Safety analysis set included all participants who received the study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 7
percentage of participants | 28.6

9. Secondary Outcome: Percentage of Participants With At Least One Treatment-Emergent Adverse Event of Special Interest (AESI)
Description: AESIs include immunogenicity/alloimmune reactions, hypersensitivity reactions, ectopic tissue formation, medication errors, tumorigenicity, and transmission of infectious agents. A treatment-emergent AESI is an AESI which occurs after exposure to study treatment.
Time Frame: Up to Week 52
Population: Safety analysis set included all participants who received the study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 7
percentage of participants | 0.0

10. Secondary Outcome: Percentage of Participants With Potentially Clinically Significant Vital Sign Values
Description: Vital signs include body temperature (oral measurement), blood pressure (systolic and diastolic, resting more than 5 minutes), and heart rate (beats per minute).
Time Frame: Up to Week 52
Population: Safety analysis set included all participants who received the study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 7
percentage of participants | 0.0

11. Secondary Outcome: Percentage of Participants With Potentially Clinically Significant Laboratory Values
Description: Laboratory parameters include hematology, biochemistry, and urinalysis.
Time Frame: Up to Week 52
Population: Safety analysis set included all participants who received the study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Darvadstrocel
Number analyzed (Participants) | 7
percentage of participants | 0.0

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: Safety analysis set included all participants who received the study treatment.
Arm/Group | Darvadstrocel
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darvadstrocel (N=7)
Anal abscess (Infections and infestations) | 1
Proctalgia (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Darvadstrocel (N=7)
Anaemia (Blood and lymphatic system disorders) | 1
Anal abscess (Infections and infestations) | 1
Anal fistula (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Influenza (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT04701411/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT04701411/SAP_001.pdf